CLINICAL TRIAL: NCT06203015
Title: The Relations Among Endotoxin, Inflammatory Cytokines, Cognitive Markers and Brain MRI Changes in Subjects With Depressive Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Vesta Steibliene, Professor, Lithuanian University of Health Sciences
Other Study IDs: DEPRINFLAMATION-Versija 3
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Major Depressive Disorder; Inflammation; Cognitive Dysfunction; Endotoxemia; Genetic Predisposition to Disease; Blood Brain Barrier Defect
Keywords: Major depressive disorder; Inflammation; Endotoxin; Cognitive dysfunction; Genetic polymorphisms; Multiparametric Magnetic Resonance Imaging; Blood Brain Barrier
MeSH Terms: conditions — Depressive Disorder, Major; Inflammation; Cognitive Dysfunction; Endotoxemia; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MDD patients: patients diagnosed with MDD (according to the WHO's [2019] International Classification of Diseases and related health problems categorization of mental disorders), diagnosed by a psychiatrist; ≥18 years old
  Interventions: Diagnostic Test: The Cambridge Neuropsychological Test Automated Battery.; Diagnostic Test: Venous blood samples; Diagnostic Test: brain MRI; Diagnostic Test: the Montgomery-Åsberg Depression Rating Scale; Other: questionnaire prepared by the researchers
- Control group: Subjects who have not been diagnosed with any mental disorder in the past year; ≥18 years old
  Interventions: Diagnostic Test: The Cambridge Neuropsychological Test Automated Battery.; Diagnostic Test: Venous blood samples; Diagnostic Test: brain MRI; Diagnostic Test: the Montgomery-Åsberg Depression Rating Scale; Other: questionnaire prepared by the researchers

INTERVENTIONS:
Diagnostic Test: The Cambridge Neuropsychological Test Automated Battery. — to determine cognitive dysfunction
Diagnostic Test: Venous blood samples — to measure levels of cytokines, endotoxin, and genetic markers.
Diagnostic Test: brain MRI — to evaluate BBB permeability to water, brain structure volumes, white matter integrity, cerebral perfusion, and neurometabolite concentrations
Diagnostic Test: the Montgomery-Åsberg Depression Rating Scale — to measure severity of depressive symptoms
Other: questionnaire prepared by the researchers — collecting sociodemographic data and information about smoking status, BMI, data on the course of MDD, past treatment, comorbid diseases, and current use of medications.

SUMMARY:
Major depressive disorder (MDD) is a chronic mental illness, with 60% lifetime risk of recurrence after the first MDD episode. Despite available treatment options for MDD, only about half to two-thirds of patients respond to first-line antidepressant treatment, and only 30% to 45% of patients achieve remission. Scholars assume that this low remission rate and high rate of treatment resistance are due to the polyetiological nature of the disease, the heterogeneity of the clinical picture of depression, and the lack of biomarkers to stratify MDD subtypes. The aetiology of MDD, although researched extensively, remains unclear. None of the known mechanisms alone explains the pathogenesis of depression, meaning that the interplay of several factors contributes to the development of MDD. Accumulated scientific evidence has supported the importance of the immune system in the etiopathogenesis of MDD. Until now, the cause of the low-grade inflammation observed in this subgroup of MDD patients has been unclear. In the proposed study, the investigators will test a new hypothesis of the immune theory of the development of MDD: the endotoxin hypothesis of neurodegeneration. This hypothesis states that endotoxin, causes or contributes to neurodegeneration. Blood plasma levels of LPS are normally low but are elevated during infections, gut inflammation, gum disease, and neurodegenerative diseases. Dysbiosis may promote increased intestinal permeability ("leaky gut"), which leads to bacterial translocation across the intestinal barrier and into the circulation, thus forming of LPS and LPS-binding protein complex, which triggers the secretion of cytokines. Data suggest that LPS-induced peripheral inflammation can activate neuroinflammation. However, it is not known whether a low-level persistent presence of LPS in the circulatory system can cause low-grade chronic neuroinflammation leading to neurodegeneration and/or symptoms of MDD. Based on existing preclinical and clinical research data, the investigators hypothesise that an increase in blood plasma endotoxin and peripheral cytokines induce BBB dysfunction, neuroinflammation and neurodegenerative processes in specific etiologically relevant structures of the brain and cause clinical manifestation of depressive symptoms and cognitive damage. In this study the investigators are also going to investigate the effects of single nucleotide polymorphisms of four genes in relation to blood plasma endotoxin and peripheral cytokines concentrations and clinical manifestation of MDD.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* signed informed consent
* patients diagnosed with MDD (according to the WHO's [2019] International Classification of Diseases and related health problems categorization of mental disorders) for MDD group.

Exclusion Criteria:

* diagnosis of other mental disorders during the past one-year period (for MDD group).
* diagnosis of any mental disorders within the past one-year period, previous suicide attempt, or current suicide risk identified in the study (for control group).
* diagnosis of somatic diseases that may affect changes in inflammatory factors in the body (for both groups)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is being conducted at the hospital of the Lithuanian University of Health Sciences Kaunas Clinics Psychiatry Clinic (inpatient department), and the Nervous System Diseases Outpatient Department.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Levels of blood plasma endotoxin and inflammatory cytokines between groups. | Day 1
  To evaluate the concentrations of blood plasma endotoxin and inflammatory cytokines among patients with MDD and in a control group. We hypothesize that an increase in blood plasma endotoxin is associated with an increase in blood inflammatory cytokines in the group of patients with MDD.
Severity and manifestation of depressive symptoms. | Day 1
  Evaluate the severity and manifestation of different depressive symptoms. We hypothesize that endotoxin and inflammatory markers are associated with specific symptoms of MDD, allowing us to identify MDD patients with a specific LPS-induced/stimulated inflammatory depression subtype.

SECONDARY OUTCOMES:
Brain MRI | Day 1
  Perform a multiparametric brain MRI assessment of depressed patients and a control group. We hypothesize that, among patients with MDD, there are changes in blood-brain barrier permeability to water, levels of neuroinflammation and perfusion, and structural neurodegenerative changes that are associated with blood plasma endotoxin and cytokine concentrations.
Cognitive dysfunction | Day 1
  Evaluate cognitive functions. We hypothesize that low-grade neuroinflammation negatively affects cognitive performance among patients with MDD.
Covariates | Day 1
  Perform a subgroup analysis on neuroinflammation markers based on individuals' BMI and smoking status.
Genetic markers | Day 1
  Determine possible genetic markers among MDD subjects in relation to blood plasma endotoxin and inflammatory cytokines concentrations that could predict a genetic predisposition to neuroinflammation, neurodegeneration and the development of MDD.

CONTACTS AND LOCATIONS:
Overall Officials: Vesta Steibliene, PhD, MD, Principal Investigator — Proffesor, Lithuanian University of Health Sciences
Locations (1):
- Psychiatry Department, Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas, Lithuania

REFERENCES:
- [Derived] Milasauskiene E, Burkauskas J, Jesmanas S, Gleizniene R, Borutaite V, Skemiene K, Vaitkiene P, Adomaitiene V, Lukosevicius S, Gradauskiene B, Brown G, Steibliene V. The links between neuroinflammation, brain structure and depressive disorder: A cross-sectional study protocol. PLoS One. 2024 Nov 20;19(11):e0311218. doi: 10.1371/journal.pone.0311218. eCollection 2024. PMID 39565757